

HIIT + Age: Effects of High-Intensity Interval Training on Functional Fitness in Older Adults

Ethical number: 2067313

ClinicalTrials.gov Identifier (NCT Number): NCT99999999 (to be updated upon

registration)

**Date of Document: April 2024** 



#### **Informed Consent Form**

Each research participant must sign this document to authorize their participation. This form will be securely stored by the principal investigator. This model is in accordance with the Declaration of Helsinki and the Oviedo Convention.

**Information:** Please read the following information carefully. If anything is unclear or incorrect, do not hesitate to request further clarification. If you agree to participate, please sign this document.

## Research Project Title: + Age + Health - HIIT

**Summary:** Aging is associated with a decline in functional fitness, compromising autonomy and quality of life. Strategies such as high-intensity interval training (HIIT) have gained attention for their positive effects on various physical parameters. This study evaluates the effectiveness of a HIIT program in improving strength, mobility, flexibility, and aerobic endurance in older adults. The results reinforce its potential as a safe and effective tool for promoting functionality and independence in the elderly population.

**Purpose:** To assess the feasibility and effectiveness of a high-intensity interval training (HIIT) program on functional fitness in older adults.

Funding: This research has not received any financial support.

**Confidentiality and Anonymity:** Researchers will obtain informed consent from all participants. This study adheres to the Declaration of Helsinki and was approved by the Ethics Committee of the Polytechnic Institute of Bragança (approval number: [2067313]).

Research Group: António Miguel Monteiro<sup>1\*</sup>, André Schneider<sup>1</sup>

**Affiliations:** <sup>1</sup>Department of Sport Sciences, Instituto Politécnico de Bragança (IPB), 5300-253 Bragança, Portugal; andrecschneider@gmail.com; mmonteiro@ipb.pt

\*Autor correspondente: mmonteiro@ipb.pt

## **Procedures and Timeline**

If you agree to participate in this study, you will be asked to undergo three assessments at different time points:

- 1. First Assessment: At the beginning of the study (baseline, week 0).
- Second Assessment: Midway through the study (~33 week).
- 3. Third Assessment: At the end of the study (~65 week).

he multicomponent training program consists of three weekly sessions. The study groups are as follows:

- Control Group: Will not undergo training but will be assessed at all the same time points.
- Intervention Group: Will participate in supervised high-intensity interval training (HIIT) sessions.

The assessments will include:

1. Functional Fitness: Tests of strength, balance, flexibility, and endurance.

#### **Participant Responsibilities**

If you agree to take part in this study, you will be required to:

- 1. Attend all scheduled assessments and training sessions (if assigned to the intervention group).
- 2. Inform the research team of any adverse events or difficulties experienced during the study.

## Withdrawal from the Study

You may withdraw your consent and leave the study at any time without penalty or consequences. If you decide to leave the study, please notify the researchers immediately.

The researchers may also terminate your participation for reasons such as:

- Failure to follow the study instructions;
- Situations where your health may be at risk;
- Study cancellation for administrative or other reasons.



# Participant Statement

| risks, and benefits. I understand that my participation is voluntary and that I may withdraw at any time. I also authorize the anonymous use of my data for scientific purposes. |
|---|
| FULL NAME: |
| Signature: |
| Researcher signature: |

I, [full name of the participant], declare that I have read and understood the terms of this document. I voluntarily agree to participate in the research project described above, after being informed about the objectives, procedures, potential

